CLINICAL TRIAL: NCT01234961
Title: Outcomes of the Work Rehabilitation Method Redesigning Daily Occupations (ReDO) - a Quasi-experimental Study Among Women With Stress-related Disorders
Brief Title: Outcome Study of the ReDO Intervention for Women With Stress-related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Principal Investigator, Mona Eklund, Professor, Lund University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAS2005_ME; 2004-0615 (Other Grant/Funding Number: Swedish Council for Working Life and Social Research)
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Adjustment Disorders; Burnout, Professional
MeSH Terms: conditions — Adjustment Disorders; Burnout, Professional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Redesigning Daily Occupations (Experimental): The ReDO intervention focuses on how people compose their everyday lives. Supporting people in how to change and modify their patterns of daily occupations is a new intervention method for people with stress-related disorders, but it has been shown to be effective in improving quality of life and self-rated health in other target groups. The basic idea is that re-structuring of an individual's lifestyle and pattern of daily occupations will lead to a healthier balance between the occupations of everyday life, and that this balance will promote wellness and improved work capacity. The program is group based and comprises 16 weeks, with sessions 2 x 2 hours per week, followed by 3-4 booster sessions.
  Interventions: Behavioral: Redesigning Daily Occupations
- Care as usual (Active Comparator): Standard rehabilitation provided by the Social Insurance Office, such as stress management, physical therapy, mindfulness training.
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Redesigning Daily Occupations — The ReDO is a 16-week group-based programme, comprising three phases. Phase I covers five weeks and has a special focus on occupational self-analysis, while Phase II, also comprising five weeks, is concentrated around goal setting and strategies for accomplishing desired changes in the patterns of everyday activities. During these ten weeks the group meets twice a week and each session lasts for 2½ hrs. Phase III consists of work placement for six weeks, if possible in relation to the woman's ordinary work but otherwise at another relevant work place. During Phase III the group meets three times (weeks two, four and six) in order to monitor the group placement. The groups are led by two licensed occupational therapists specifically trained for the ReDO programme.
  Arms: Redesigning Daily Occupations
Other: Care as usual — The CAU group gets follow-ups by an officer at the Social Insurance Office, including contacts with the employer, but the additional support varies largely, from receiving relevant medical care, if any, to physical therapy and to more comprehensive rehabilitation programmes.
  Arms: Care as usual

SUMMARY:
This project evaluates the outcomes of a work rehabilitation program, Redesigning Daily Occupations (ReDO), for women with stress-related disorders. The ReDO intervention focuses on how people compose their everyday lives. The basic idea is that re-structuring of an individual's lifestyle and pattern of daily occupations will lead to a healthier balance between the occupations of everyday life, and that this balance will promote wellness and increased work capacity. The program is group based and comprises 16 weeks.

The aim is to evaluate ReDO for women with stress-related disorders. The project, which covers the time period from entering the program to a 12-month follow-up, is a quasi-experimental study. 42 women who entered the program and fitted the selection criteria were included. A matched comparison group was selected among those clients at the Social Insurance Office who get "care-as-usual" (CAU). Both groups are followed prospectively and are compared regarding return to work, sick leave, and different aspects of health and well-being. The hypothesis is that the ReDO group will improve more than the CAU group in all these respects.

DETAILED DESCRIPTION:
This project is about developing and evaluating a novel work rehabilitation program, Redesigning Daily Occupations (ReDO), for women with stress-related disorders. It is a co-operation project between Lund University, the Social Insurance Office, and the health care services of the County of Halland. The ReDO intervention focuses on how people compose their everyday lives. Supporting people in how to change and modify their patterns of daily occupations is a new intervention method for people with stress-related disorders, but it has been shown to be effective in improving quality of life and self-rated health in other target groups. The basic idea is that re-structuring of an individual's lifestyle and pattern of daily occupations will lead to a healthier balance between the occupations of everyday life, and that this balance will promote wellness and increased work capacity. The program is group based and comprises 16 weeks, with sessions 2 x 2 hours per week, followed by 3-4 booster sessions.

The aim of the research project is to evaluate the outcomes of ReDO for women with stress-related disorders. The hypothesis is that the ReDO group will improve more than a comparison group receiving "care-as-usual" (CAU) regarding return to work, sick leave, and different aspects of health and well-being. group in all these respects.

The project is a quasi-experimental study. It covers the time period from entering the program to a 12-month follow-up. According to initial plans, the first 50 women who entered the ReDO program and fitted the selection criteria would be included. A power analysis indicated that 40 individuals in each group were needed to detect a medium effect size (of 0.6) with 80% power at p<.05. Forty-two women were actually recruited to the ReDO intervention. A matched comparison group was selected among those clients at the Social Insurance Office who get (CAU). The match was made on specific diagnosis, age, family situation (civil status and number of children), type of occupation and duration of sick leave. Thus, in all 84 women take part in the project. The data consist of registry information from the Social Insurance Office (SIO) and questionnaires targeting socio-demographics, perceived stress, and different aspects of health and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adjustment disorder or Burnout
* Being on sick-leave for > 2 months (full time or part time)
* Having an employment

Exclusion Criteria:

* Other main diagnosis than Adjustment disorder or Burnout

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Return to work | baseline
Return to work | 12-months

SECONDARY OUTCOMES:
Perceived stress | baseline
Perceived stress | 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Mona Eklund, Principal Investigator — Department of Health Sciences, Lund University
Locations (1):
- Halland County Concil primary health care services, Halmstad, Sweden

REFERENCES:
- [Derived] Eklund M, Erlandsson LK, Wastberg BA. A longitudinal study of the working relationship and return to work: perceptions by clients and occupational therapists in primary health care. BMC Fam Pract. 2015 Apr 10;16:46. doi: 10.1186/s12875-015-0258-1. PMID 25887461
- See also: Link to the home page of the research group (currently under construction) — http://www.med.lu.se/english/hvs/activity_and_health